CLINICAL TRIAL: NCT04445272
Title: A Multicentre, Open-label Clinical Trial to Evaluate the Effectiveness and Safety of Intravenous Tocilizumab for Treating Patients With COVID-19 Pneumonia: the BREATH-19 Study
Brief Title: Clinical Trial to Evaluate the Effectiveness and Safety of Tocilizumab for Treating Patients With COVID-19 Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: Roche Pharma AG (Industry); Dynamic Science S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BREATH-19 (FSG011-20)
Record Dates: First submitted 2020-06-13; First posted 2020-06-24 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Phase II, one-arm, open label, multicentre study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tocilizumab (Experimental): Patients will receive IV tocilizumab as per clinical practice and at the discretion of treating investigator, following the posology indicated in the SmPC, or the recommendations proposed by the Spanish Ministry of Health:
  The recommended posology by the SmPC is 8 mg per kg in patients weighing greater than or equal to 30 kg or 12 mg per kg in patients weighing less than 30 kg. If no clinical improvement in the signs and symptoms up to 3 additional doses of tocilizumab may be administered. The interval between consecutive doses should be at least 8 hours.
  The recommendations of the Spanish Ministry of Health:
  Patients more than 80 kg: first dose 600 mg; second dose 600 mg. Patients less than 80 kg: first dose 600 mg; second dose 400 mg.
  A third dose might be considered 16 to 24 hours after if: fever persists or a worsening of the laboratory parameters
  Given the exceptionality of the situation modification of doses according to the physician experience will be allowed.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Treatment with Tocilizumab

SUMMARY:
At present, no treatment has been approved for COVID-19. However, in light of the increased interest on using the anti-cytokine therapy targeting IL-6 tocilizumab in COVID-19 infected patients due to its potential benefit, the Spanish Agency for Medicine and Health Products (Agencia Española de Medicamentos y Productos Sanitarios, AEMPS) have initiated the controlled distribution of the drug. Tocilizumab is indeed proposed as a potential treatment for severe COVID-19 in Spain. Based on the positive results of tocilizumab in the treatment of COVID-19 patients and the experience of tocilizumab in inducing rapid reversal of CSS in other pathologies several clinical trials and observational studies are being conducted to assess the effectiveness and safety of tocilizumab in COVID-19 patients. Further studies with a large sample size are required to confirm the effectiveness of tocilizumab in patients with COVID-19 pneumonia.

The need for the management of severe COVID-19 disease is imperative, and every effort should be made to collect relevant clinical outcomes. The aim of the present study is to evaluate the effectiveness of IV tocilizumab in treating patients with COVID-19 pneumonia who are currently hospitalized or admitted to ICU by describing improvement of respiratory function and mortality rate. This large real-world cohort therefore provides a unique opportunity to study this potential medicine during the current emergency situation, and support the findings from other ongoing clinical trials and observational studies, such as the Roche-sponsored Phase III study that is planned to start early April.

DETAILED DESCRIPTION:
Cytokine storm syndrome (CSS) is caused by the excessive release of cytokines during an exaggerated immune response. CSS can be triggered by infections or therapeutic interventions, being more severe depending on the degree and duration of immune activation. CSS is as a significant on-target side-effect of chimeric antigen receptor (CAR) T-cell therapies, which have been subject to assessment for the treatment of haematological malignancies. Tocilizumab (intravenous, IV) is indicated for the treatment of chimeric antigen receptor CAR T cell-induced severe or life-threatening CSS.

Based on the experience with tocilizumab in the CSS, and that some patients infected with SARS-CoV-2 can develop CSS, leading to potentially fatal damage to lung tissue, the drug is being investigated in China and Italy, and clinical trials are being conducted/planned in these and several other countries. Real-word experience with tocilizumab IV have shown that in a substantial proportion of COVID-19 patients with severe pneumonia, fever returned to normal and respiratory function based on oxygen intake and lung opacities improved remarkably. Laboratory parameters such as C-reactive protein (CRP) that seem to be increased in patients infected decreased significantly with tocilizumab, and lymphocytes levels also returned to normal.

All these findings have led the Spanish Agency for Medicine and Health Products (AEMPS) to initiate the controlled distribution of tocilizumab IV, in light of the increased interest on the anti-cytokine therapy targeting IL-6 in COVID-19 infected patients. Therefore, tocilizumab might be among the therapeutic armamentarium for preventing the fatal consequences of acute respiratory and multi organ failure in around 20% of the COVID-19 infected patients.

The aim of the present study is to evaluate the effectiveness and safety of IV tocilizumab in patients with COVID-19 severe pneumonia who are currently hospitalized or admitted to ICU. This large real-world cohort provides a unique opportunity to study a potential medicine during the current emergency situation, and support the findings from the Roche-sponsored Phase III study that is planned to start in early April.

ELIGIBILITY:
Inclusion Criteria:

* Provide oral informed consent to participate in this study.
* At least 18 years of age.
* Diagnosed with COVID-19 pneumonia by RT-PCR.
* Have received the first dose of tocilizumab a maximum of two days before the inclusion or is candidate for tocilizumab treatment
* Hospitalized or admitted to ICU

Exclusion Criteria:

* The patient has any other medical condition or is receiving concomitant medication that could, in the opinion of the investigator, compromise the patient's safety or collected data
* Known severe allergic reactions to tocilizumab or other monoclonal antibodies
* Active acute and severe infections, including tuberculosis infection
* Pregnant or breastfeeding, or positive pregnancy test in a pre-dose examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
To calulate the time of intubation | through study completion, and average of 1 month
  Calculate the mean time of intubation
To calculate the time with oxygen therapy | through study completion, and average of 1 month
  Calculate the mean time with oxygen therapy
To calculate the time with Non-invasive mechanical ventilation | through study completion, and average of 1 month
  Calculate the mean time with Non-invasive mechanical ventilation
To evaluate mortality rate | through study completion, and average of 1 month
  Number of patients deaths of the total of patients included

SECONDARY OUTCOMES:
To calculate respiratory function parameters | through study completion, and average of 1 month
  To calculate the mean ofPaO2/FiO2
To calculate respiratory function parameters | through study completion, and average of 1 month
  To calculate the mean of levels of oxygen saturation
To calculate respiratory function parameters | through study completion, and average of 1 month
  To calculate the mean of SaO2/FiO2
To evaluate radiological lung extension | through study completion, and average of 1 month
  Evaluate the lung extension of pneumonia
To evaluate radiological evolution | through study completion, and average of 1 month
  Evaluate the type of lung affection
To describe the duration of hospitalization and ICU use | through study completion, and average of 1 month
  Days of hospitalization in survivors and/or days at ICU throughout the study
To evaluate the requirement of additional organ support | through study completion, and average of 1 month
  Percentage of patients with extracorporeal membrane oxygenation
To evaluate the requirement of additional organ support | through study completion, and average of 1 month
  Percentage of patients with molecular adsorbent recirculating system
To evaluate the requirement of additional organ support | through study completion, and average of 1 month
  Percentage of patients with dialysis
To evaluate the requirement of additional organ support | through study completion, and average of 1 month
  Percentage of patients with other support therapy
To evaluate the effect of IV tocilizumab on the serum levels of inflammatory markers | through study completion, and average of 1 month
  Analyze the levels of IL-6
To calculate the number of adverse events in patients with COVID-19 pneumonia treated with Tocilizumab | through study completion, and average of 1 month
  Incidence of adverse events
To calculate the number of adverse events in patients with COVID-19 pneumonia treated with Tocilizumab | through study completion, and average of 1 month
  Incidence of adverse events by dose of Tocilizumab
To assess time to reverse-transcriptase polymerase chain reaction (RT-PCR) virus negativity | through study completion, and average of 1 month
  To evaluate the time to RT-PCR virus negativity
To evaluate the effect of IV tocilizumab on the serum levels of inflammatory | through study completion, and average of 1 month
  Analyze the levels of CRP
To evaluate the effect of IV tocilizumab on the serum levels of inflammatory | through study completion, and average of 1 month
  Analyze the levels of procalcitonin (PCT)
To evaluate the effect of IV tocilizumab on the serum levels of inflammatory | through study completion, and average of 1 month
  Analyze the levels of ID-dimer
To evaluate the effect of IV tocilizumab on the serum levels of inflammatory | through study completion, and average of 1 month
  Analyze the levels of ferritin
To calculate the number of serious adverse events in patients with COVID-19 pneumonia treated with Tocilizumab | through study completion, and average of 1 month
  Indicende of serious adverse events
To calculate the number of serious adverse events in patients with COVID-19 pneumonia treated with Tocilizumab | through study completion, and average of 1 month
  Indicende of serious adverse events based on dose of Tocilizumab
To calculate the number of adverse events of special interest in patients with COVID-19 pneumonia treated with Tocilizumab | through study completion, and average of 1 month
  Indicende of adverse events of special interest based on dose of Tocilizumab
To evaluate mortality rate | through study completion, and average of 1 month
  Number of patients deaths of the total of patients included based on dose of Tocilizumab
To evaluate respiratory function | through study completion, and average of 1 month
  Time with intubation, oxygen therapy and Non-invasive mechanical ventilation based on dose of Tocilizumab
To evaluate mortality rate | through study completion, and average of 1 month
  Number of patients deaths of the total of patients included based on severity of disease at the start of the study treatment
To evaluate mortality rate | through study completion, and average of 1 month
  Number of patients deaths of the total of patients included based on presence of cytokine storm syndrome at the start of treatment
To evaluate respiratory function | through study completion, and average of 1 month
  Time with intubation, oxygen therapy and Non-invasive mechanical ventilation based on severity of disease at the start of the study treatment
To evaluate respiratory function | through study completion, and average of 1 month
  Time with intubation, oxygen therapy and Non-invasive mechanical ventilation based on presence of cytokine storm syndrome at the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jose Antonio Pérez Molina, Principal Investigator — Hospital Universitario Ramón y Cajal
Locations (42):
- Spain (42):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Sant Joan de Déu de Manresa, Manresa, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Universitario de Galdakao, Galdakao, Bizkaia
  - Hospital Universitario Marqués Valdecilla, Santander, Cantabria
  - Hospital Público General del Tomelloso, Tomelloso, Ciudad Real
  - Hospital Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Rey Juan Carlos, Móstoles, Madrid
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario de Cabueñes, Gijón, Principality of Asturias
  - Hospital Nuestra Señora del Prado, Talavera de la Reina, Toledo
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital Infanta Cristina, Badajoz
  - Hospital Clínic i Provincial Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Dr. Josep Trueta, Girona
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitario Salamanca, Salamanca
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Poliectenic La Fe, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maude SL, Barrett D, Teachey DT, Grupp SA. Managing cytokine release syndrome associated with novel T cell-engaging therapies. Cancer J. 2014 Mar-Apr;20(2):119-22. doi: 10.1097/PPO.0000000000000035. PMID 24667956